CLINICAL TRIAL: NCT04811430
Title: Comparative Effectiveness, Efficiency, and Emergency Department Nurse Preference Between 2 Methods of Visualization for Midline Catheter Insertion: A Pilot Study
Brief Title: Efficiency, and Emergency Department Nurse Preference Between 2 Methods of Visualization: A Pilot Study
Status: Completed | Type: Observational
Sponsor: Becton, Dickinson and Company (Industry)
Responsible Party: Sponsor
Other Study IDs: P88008.0
Record Dates: First submitted 2021-03-19; First posted 2021-03-23 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Catheter Related Complication
Keywords: Visualization; Needle Guidance; Midline Catheter; Emergency Department Nurse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Randomized Traditional: Randomized to traditional ultrasound guided peripheral insertion placement vs placement with Cue needle tracking technology
  Interventions: Device: Randomized Traditional; Device: Cue(TM) Needle Tracking Technology
- Radomized Cue Needle Tracking technology: Randomized to traditional ultrasound guided peripheral insertion placement vs placement with Cue needle tracking technology
  Interventions: Device: Randomized Traditional; Device: Cue(TM) Needle Tracking Technology

INTERVENTIONS:
Device: Randomized Traditional — Traditional ultrasound guidance was utilized to insert Midlines on simulated veins blocks not live patients
  Other Names: Randomized Traditional Ultrasound method
Device: Cue(TM) Needle Tracking Technology — Cue(TM) Needle Tracking Technology with real time needle tip tracking is used to assist ultrasound guided midline insertions on simulated veins blocks not live patients

SUMMARY:
The purpose of this study was to assess the impact of a continuous needle tracking system on the accuracy, speed, and quality of ultrasound-guided peripheral venous catheter insertion.

DETAILED DESCRIPTION:
A pilot study using simulated tissue was conducted with 49 US-based emergency department nurses to compare insertion of a midline catheter using traditional ultrasound guidance versus an advanced needle-tracking technology along with traditional ultrasound guidance.

ELIGIBILITY:
Inclusion Criteria:

* US-based emergency department nurse who have placed 10 peripheral intravenous catheters in the past 60 days
* have placed less than or equal to 15 ultrasound-assisted vascular access devices in the past 60 days and have been practicing ultrasound-assisted vascular access no more than 18 months

Exclusion Criteria:

* Nurses that don't meet that predetermined inclusion criteria

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Emergency Department and Critical Care Nurses
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2019-10-14 (Actual); Study Completion 2019-10-15 (Actual)

PRIMARY OUTCOMES:
Insertion Success | 1 hour
  Number of attempts required to properly place a needle tip in the simulated vessel
Insertion Time | 1 hour
  Time required to successfully insert a needle tip into a simulated vessel
Backwalling Events | 1 hour
  Events where the needle fully transects the simulated blood vessel during the inserting of the needle tip into a simulated vessel
Needle redirects | 1 hour
  Lateral movement and deflection of the needle tip during insertion into a simulated vessel
Accuracy of Needle Placement | 1 hour
  Accuracy of needle placement as indicated by the lateral distance from a target

SECONDARY OUTCOMES:
Self-reported subjective measurements | 1 hour
  Post-study questions were used to assess confidence during insertion with Cue needle tracking system (likert), confidence when insertion with traditional ultrasound techniques (likert), preference between the cue needle tracking system and the standard of care

CONTACTS AND LOCATIONS:
Locations (1):
- Austin Convention Center, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No